CLINICAL TRIAL: NCT06955143
Title: A Study on Integrated Multi-Omics and Multi-Factor Analysis of Peripheral Blood in Patients With Acute Coronary Syndrome
Brief Title: A Study on the Peripheral Blood in Patients With Acute Coronary Syndrome
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: The Central Hospital of Lishui City (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-06-218
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Acute Coronary Syndrome; Chronic Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ACS: those with a condition of Acute Coronary Syndrome
- Control: patients without coronary artery disease, valvular heart disease, structural heart disease, or any other kind of cardiomyopathy
- CCS: those with a condition of Chronic Coronary Syndrome

SUMMARY:
The goal of this study is to conduct analyses the changes of cell growth factors, inflammatory factors, metabolites, plasma proteome, etc. in the blood of patients with ACS (acute coronary syndrome), as well as their correlations with the disease prognosis, based on multi-omics or other related research methods. The main questions it aims to answer are:

The growth factors that have significant changes in the peripheral blood of the ACS population, especially fibroblast growth factors? Inflammatory factors and chemokines related to the onset of ACS? The metabolites and proteins that are significantly altered in the peripheral blood after the onset of ACS? Researchers will compare ACS population to CCS (Chronic Coronary Syndrome) population, and control group (patients without coronary artery stenosis, valvular heart disease, structural heart disease, or any other kind of cardiomyopathy).The peripheral venous blood from the participants will be collected within 24 hours after their admission to the hospital.

ELIGIBILITY:
Inclusion Criteria:

For ACS group STEMI

* cTn>99th ULN or CK-MB>99th ULN
* ST-segment elevation with a convex upward morphology
* in conjunction with one or more of the following conditions: persistent ischemic chest pain; echocardiographic evidence of abnormal segmental ventricular wall motion; or abnormal coronary angiography findings.

NSTEMI

* cTn>99th ULN or CK-MB>99th ULN
* accompanied by one or more of the following situations: persistent ischemic chest pain; new ST-segment depression or low and inverted T waves; echocardiography showing segmental ventricular wall motion abnormalities; abnormal coronary angiography.

UA

* cTn normal
* ischemic chest pain with an electrocardiogram showing transient ST-segment depression or flattened and inverted T waves
* evidence of coronary artery stenosis (e.g., CTA demonstrating ≥ 50% stenosis) For CCS group
* Clinical Diagnosis Consistent with CCS Categories, meet any one of the following clinical scenarios: Stable Angina Pectoris, Ischemic Cardiomyopathy, Post-ACS Stable Phase, Long-Term CAD Management, Vasospastic or Microvascular Disease, Asymptomatic CAD
* Laboratory and Imaging Confirmation: Resting ECG without ST-segment elevation or dynamic changes (excluding ACS), cTn normal or stable (no acute myocardial injury), ≥50% luminal stenosis in ≥1 epicardial coronary artery For control group
* Patients without coronary artery stenosis, valvular heart disease, structural heart disease, or any other kind of cardiomyopathy

Exclusion Criteria:

* Lactating or pregnant women
* Patients with malignant neoplasms
* Severe hepatic/renal dysfunction
* Severe hematological disorders
* Autoimmune diseases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who presented to Lishui Central Hospital (Fifth Affiliated Hospital of Wenzhou Medical University) due to cardiac discomfort or other related symptoms were consecutively enrolled in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
circulating fibroblast growth factors (FGFs) levels | within 24 hours of admission to the hospital
  examining the circulating fibroblast growth factors levels in the peripheral venous blood of the participants
circulating inflammatory cytokines levels | within 24 hours of admission to the hospital
  examining the circulating inflammatory cytokines levels in the peripheral venous blood of the participants
circulating chemokines levels | within 24 hours of admission to the hospital
  examining the circulating chemokines levels in the peripheral venous blood of the participants
circulating Cytochrome C level | within 24 hours of admission to the hospita
  examining the circulating cytochrome c levels in the peripheral venous blood of the participants
circulating mitochondrial DNA levels | within 24 hours of admission to the hospital
  examining the circulating mitochondrial DNA levels in the peripheral venous blood of the participants
circulating malondialdehyde levels | within 24 hours of admission to the hospital
  examining the circulating malondialdehyde levels in the peripheral venous blood of the participants

SECONDARY OUTCOMES:
the relationship between FGFs/inflammatory cytokines/chemokines and troponin I (TnI) | within 24 hours of admission to the hospital
  performed correlation analyses between the circulating levels of FGFs/inflammatory cytokines/chemokines and TnI
the relationship between FGFs/inflammatory cytokines/chemokines and brain natriuretic peptide (BNP) | within 24 hours of admission to the hospital
  performed correlation analyses between the circulating levels of FGFs/inflammatory cytokines/chemokines and BNP
the relationship between FGFs/inflammatory cytokines/chemokines and lactate dehydrogenase (LDH) | within 24 hours of admission to the hospital
  performed correlation analyses between the circulating levels of FGFs/inflammatory cytokines/chemokines and LDH
the relationship between FGFs/inflammatory cytokines/chemokines and left ventricular ejection fraction (LVEF) | within 24 hours of admission to the hospital
  performed correlation analyses between the circulating levels of FGFs/inflammatory cytokines/chemokines and LVEF
the relationship between FGFs/inflammatory cytokines/chemokines and mitochondrial DNA (mitoDNA) | within 24 hours of admission to the hospital
  performed correlation analyses between the circulating levels of FGFs/inflammatory cytokines/chemokines and mitochondrial DNA contents
the relationship between FGFs/inflammatory cytokines/chemokines and cytochrome c | within 24 hours of admission to the hospital
  performed correlation analyses between the circulating levels of FGFs/inflammatory cytokines/chemokines and cytochrome c
the relationship between FGFs/inflammatory cytokines/chemokines and malondialdehyde | within 24 hours of admission to the hospital
  performed correlation analyses between the circulating levels of FGFs/inflammatory cytokines/chemokines and malondialdehyde

CONTACTS AND LOCATIONS:
Locations (1):
- Lishui Central Hospital, Lishui, Zhejiang, China